CLINICAL TRIAL: NCT00739934
Title: An Open-Label, Intravenous To Oral Switch, Multiple Dose Study To Evaluate The Pharmacokinetics, Safety And Tolerability Of Voriconazole In Immunocompromised Children Aged 2 To <12 Years Who Are At High Risk For Systemic Fungal Infection
Brief Title: Study Of The Pharmacokinetics And Safety Of Voriconazole In Children 2 To 11 Years Old Who Are At High Risk For Systemic Fungal Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1501088
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Candidiasis; Candidemia
Keywords: Open-Label; Pharmacokinetics; Intravenous to oral switch; Safety; Voriconazole; Immunocompromise; Children; High Risk For Systemic Fungal Infection.
MeSH Terms: conditions — Candidiasis; Candidemia | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children aged 2 to <12 years (Experimental): Immunocompromised children aged 2 to <12 years who are at high risk for systemic fungal infection.
  Interventions: Drug: voriconazole (Vfend)

INTERVENTIONS:
Drug: voriconazole (Vfend) — Study Days 1 to 7: IV voriconazole 7 mg/kg q12h. Study Days 8 to 14: Oral voriconazole (POS) 200 mg q12h
  Notes:
  1. If unable to switch to oral medication on Day 8, subjects can continue with IV treatment up to Day 20 before switching to oral dose.
  2. Only morning oral dose will be given on Day 14 (or the seventh day of oral dosing if IV regimen is extended). However, if clinically indicated, voriconazole treatment may be continued up to Day 30.
  (IV = Intravenous; POS = Powder for oral suspension)
  Other Names: UK-109,496; Vfend; voriconazole

SUMMARY:
In this study we will measure the concentration of the drug called voriconazole which is used to fight infections caused by fungus in children who usually are cancer patients and have their immune system down. Since we know the dose in adults, and we think we know the matching doses in the young patients ages 2 to 12 years old, we will compare the amount of drug that goes into the system with what we know works in adults. We give the drug by a needle directly into the blood, then few days later we stop that and give the drug by mouth. Meanwhile, we draw a little bit of blood at certain times to measure the drug in it.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 2 to <12 years of age.
* Require treatment for the prevention of systemic fungal infection.
* Expected to develop neutropenia (ANC <500 cells/μL) lasting more than 10 days following chemotherapy.
* Anticipated to live for more than 3 months.

Exclusion Criteria:

* Evidence of any clinically significant liver or renal function or other abnormalities such as cardiac arrhythmia, hypokalemia, hypomagnesemia or hypocalcemia.
* Documented bacterial or viral infection not responding to appropriate treatment.
* Hypersensitivity to or severe intolerance of azole antifungal agents.
* Receiving other azoles or drugs that is are prohibited in the voriconazole label or associated.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501088&StudyName=Study%20Of%20The%20Pharmacokinetics%20And%20Safety%20Of%20Voriconazole%20In%20Children%202%20To%2011%20Years%20Old%20Who%20Are%20At%20High%20Risk%20For%20Systemic%20Fungal%20

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Voriconazole intravenous (IV) multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Days 1 to 7 (up to Day 20 or more if clinically indicated). The oral maintenance dosing regimen (200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Period: Voriconazole IV
Arm/Group | All Participants
Started | 40
Completed | 34
Not Completed | 6
Not completed — Adverse Event | 6
Period: Voriconazole Oral
Arm/Group | All Participants
Started | 34
Completed | 31
Not Completed | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Voriconazole IV multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Days 1 to 7 (up to Day 20 or more if clinically indicated). The oral maintenance dosing regimen (200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Customized [Number; unit: Participants]
  2 to <6 years | 24
  6 to <12 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve Over Dosing Interval at Steady State (AUC12,ss) Following IV Administration
Description: AUC12,ss = Area under the plasma concentration-time profile from time zero (predose) to twelve hours at steady-state. AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 7 (up to Day 20 or more) at predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: Intent-to treat (ITT) population of participants who had completed pharmacokinetic (PK) blood sampling for at least one day. N = number of participants with analyzable data.
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole IV: Voriconazole IV multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Days 2 to 7 (up to Day 20 or more if clinically indicated).
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 36
μg*h/mL | 21.42 (35.05)

2. Primary Outcome: Peak Plasma Concentration at Steady State (Cmax,ss) Following IV Administration
Time Frame: Day 7 (up to Day 20 or more) at predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: ITT population of participants who had completed PK blood sampling for at least one day. N = number of participants with analyzable data.
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 36
μg/mL | 4.26 (3.73)

3. Primary Outcome: Time to Reach Cmax (Tmax) Following IV Administration
Time Frame: Day 7 (up to Day 20 or more) at predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 36
hours | 2.30 [1.00 to 4.07]

4. Primary Outcome: AUC12,ss Following Oral Administration
Description: as for outcome 1
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole Oral: Voriconazole oral dose (200 mg) was administered in the morning and evening following voriconazole IV and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
μg*h/mL | 18.64 (50.63)

5. Primary Outcome: Cmax,ss Following Oral Administration
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
μg/mL | 3.62 (4.66)

6. Primary Outcome: Tmax Following Oral Administration
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
hours | 1.07 [0.73 to 8.03]

7. Secondary Outcome: AUC12 Following IV Loading Dose
Description: AUC12 = Area under the plasma concentration-time profile from time zero (predose) to twelve hours. AUC12 was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 1 predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole IV: Voriconazole IV multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Day 1.
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 33
μg*h/mL | 7.85 (6.71)

8. Secondary Outcome: Cmax Following an IV Loading Dose
Time Frame: Day 1 predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 33
μg/mL | 2.15 (1.10)

9. Secondary Outcome: Tmax Following an IV Loading Dose
Time Frame: Day 1 predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 33
hours | 2.30 [1.72 to 4.08]

10. Secondary Outcome: Trough Concentrations (Cmin)
Time Frame: Day 7 (up to Day 20 or more) for IV; Day 7 (or later) for oral at predose
Population: ITT population of participants who had completed PK blood sampling for at least one day. N = number of participants with analyzable data; n = number of participants who contributed to data.
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Groups:
- All Treatments: Voriconazole IV multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Days 1 to 7 (up to Day 20 or more if clinically indicated). The oral maintenance dosing regimen (200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | All Treatments
Number analyzed (Participants) | 36
μg/mL
  IV Day 7 (up to Day 20) (n=36) | 0.61 (2.56)
  Oral Day 7 (up to Day 30) (n=32) | 0.52 (3.32)

11. Secondary Outcome: AUC12,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Description: as for outcome 1
Time Frame: Days 1 and 7 (up to Day 20 or more) predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole IV: Voriconazole IV multiple dose (7 mg/kg once every 12 hours) was administered in the morning and evening on Days 1 to 7 (up to Day 20 or more if clinically indicated).
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 39
μg*h/mL
  Day 1 | 20.98 (8.05)
  Day 7 (up to Day 20) | 41.95 (14.30)

12. Secondary Outcome: Cmax,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Time Frame: Days 1 and 7 (up to Day 20 or more) predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 39
μg/mL
  Day 1 | 2.97 (0.94)
  Day 7 (up to Day 20) | 4.47 (1.44)

13. Secondary Outcome: Tmax of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Description: Zero Tmax refers to the highest concentration observed for one participant at predose. The profile of the metabolite is relatively flat, which could result in slight variation in sample collection or assay process.
Time Frame: Days 1 and 7 (up to Day 20 or more) predose, 60 and 138 minutes, 4, 6, 8 and 12 hours postdose
Population: ITT population of participants who had completed PK blood sampling for at least one day. N=number of participants with analyzable data.
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 39
hours
  Day 1 | 4.00 [1.72 to 8.00]
  Day 7 (up to Day 20) | 4.00 [0.00 to 12.05]

14. Secondary Outcome: AUC12,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Description: as for outcome 1
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
μg*h/mL | 51.65 (27.88)

15. Secondary Outcome: Cmax,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
μg/mL | 5.62 (2.54)

16. Secondary Outcome: Tmax of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 7 (or later) predose, 1, 2, 4, 6, 8 and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 33
hours | 3.97 [0.92 to 8.03]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Voriconazole Oral: Voriconazole oral maintenance dosing regimen (200 mg every 12 hours) was administered following voriconazole IV in the morning and evening and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | Voriconazole IV | Voriconazole Oral
Serious Adverse Events (participants affected / at risk) | 6/40 | 13/34
Other Adverse Events (participants affected / at risk) | 39/40 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole IV (N=40) | Voriconazole Oral (N=34)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Catheter related complication (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 5
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 0 | 1
Device migration (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Cytomegalovirus test (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole IV (N=40) | Voriconazole Oral (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemolysis (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 2
Dilatation ventricular (Cardiac disorders) | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 3 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Factor VII deficiency (Congenital, familial and genetic disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
Cushingoid (Endocrine disorders) | 2 | 1
Astigmatism (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 0 | 1
Colour blindness acquired (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 2
Dry eye (Eye disorders) | 3 | 1
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Lacrimation decreased (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 6
Oral disorder (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 2 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4
Catheter related complication (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 2
Face oedema (General disorders) | 1 | 1
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 3
Gravitational oedema (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 3
Localised oedema (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 20 | 11
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 7 | 4
Pyrexia (General disorders) | 15 | 11
Suprapubic pain (General disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 3 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 4
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Engraftment syndrome (Immune system disorders) | 4 | 2
Graft versus host disease (Immune system disorders) | 3 | 4
Hypersensitivity (Immune system disorders) | 1 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 0 | 2
Candidiasis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 3
Cytomegalovirus viraemia (Infections and infestations) | 1 | 3
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis adenovirus (Infections and infestations) | 2 | 2
Herpes virus infection (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 4
Paronychia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 3 | 4
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1
Urinary tract infection viral (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Viral rhinitis (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Graft complication (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 6 | 8
Aspartate aminotransferase increased (Investigations) | 5 | 7
Bacteria blood identified (Investigations) | 1 | 0
Bacteria stool identified (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 2 | 3
Blood creatinine increased (Investigations) | 2 | 1
Blood immunoglobulin G decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 3 | 0
CSF virus identified (Investigations) | 0 | 1
Chest X-ray abnormal (Investigations) | 1 | 1
Clostridium difficile toxin test positive (Investigations) | 0 | 1
Cytomegalovirus test positive (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 5
Heart rate increased (Investigations) | 0 | 1
Hepatic enzyme decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 3 | 4
Human herpes virus 6 serology positive (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 4 | 3
Transaminases increased (Investigations) | 1 | 1
Urine cytomegalovirus (Investigations) | 1 | 1
Urine output decreased (Investigations) | 3 | 2
Virus urine test positive (Investigations) | 2 | 2
Visual tracking test abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 8 | 4
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Malignant mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Lethargy (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Staring (Psychiatric disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 2
Dysuria (Psychiatric disorders) | 4 | 6
Glycosuria (Psychiatric disorders) | 1 | 1
Haematuria (Psychiatric disorders) | 3 | 4
Oliguria (Psychiatric disorders) | 1 | 2
Pyelocaliectasis (Psychiatric disorders) | 1 | 0
Renal impairment (Psychiatric disorders) | 1 | 0
Urethral pain (Psychiatric disorders) | 0 | 1
Genital erythema (Reproductive system and breast disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 10
Rash (Skin and subcutaneous tissue disorders) | 8 | 9
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 13 | 10
Hypotension (Vascular disorders) | 2 | 1
Venoocclusive disease (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.